CLINICAL TRIAL: NCT07283276
Title: Effect of Adding Functional Core Stability Training or Cognitive Training on Balance and Postural Control in Rehabilitation of Chronic Ankle Instability
Brief Title: Effect of Functional Core Stability Training or Cognitive Training on Balance and Postural Control in Chronic Ankle Instability
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Manar Mahmoud Mohamed, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Manar-PHD
Record Dates: First submitted 2025-12-02; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Cognitive Training; Functional Core Stability Training; Balance; Distorted; Postural Control; Chronic Ankle Instability
MeSH Terms: interventions — Exercise; Cognitive Training

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- core stability (Experimental): they will receive traditional program plus functional core stability exercise
  Interventions: Other: strengthening exercises; Other: Balance training; Other: Functional core training; Other: Spinal motor control (stabilization) exercises
- cognitive training (Experimental): they will receive traditional program plus cognitive training
  Interventions: Other: strengthening exercises; Other: Balance training; Other: Cognitive training
- Core stability and cognitive training (Active Comparator): they will receive traditional program plus functional core training plus cognitive training
  Interventions: Other: strengthening exercises; Other: Balance training; Other: Functional core training; Other: Spinal motor control (stabilization) exercises; Other: Cognitive training

INTERVENTIONS:
Other: strengthening exercises — Stretch the gastrocnemius and soleus muscles for 30 seconds with 3 repetitions. Strengthen all ankle muscles using TheraBand resistance for various movements (dorsiflexion, plantar flexion, inversion, and eversion) and combined movements for 3 sets of 10 repetitions, three sessions weekly for two months. The training program includes progression from seated to standing for stretching and single-limb for bipedal calf raises.
Other: Balance training — Challenging disc training, utilized in balance studies, begins with participants standing with slightly bent knees. The dynamic balance training comprises 9 protocols focused on tracking a moving red circular target zone using a green point cursor that represents the center of pressure. Participants shift their body weight in various directions with visual feedback on a computer screen. Over 8 weeks, participants complete 16 sessions, each lasting 20 seconds with 7 seconds of rest in between. The time spent correctly tracking the target is measured and analyzed across all protocols.
Other: Functional core training — Participants will receive functional core motor control (stabilization) exercise and the traditional program (consisting of stretching protocol, strengthening of all ankle muscles, and balance activities) 3 sessions per week for 2 months.
  Arms: Core stability and cognitive training; core stability
Other: Spinal motor control (stabilization) exercises — The training program consists of three phases:
  1. **Cognitive Phase (Weeks 1-2):** Focuses on isolating the transversus abdominis and multifidus muscles using a biofeedback pressure device. Exercises involve isometric contractions with 10-second holds, repeated four times daily.
  2. **Associative Phase (Weeks 3-4):** Introduces less stable exercises (e.g., quadruped and standing positions) aimed at enhancing spine neutrality.
  3. **Automatic Phase (Weeks 5-8):** Involves dynamic movements that integrate spine control with extremity movements. Key exercises include lunges with a medicine ball, squats, and various plank variations, emphasizing co-contraction of core muscles for stability during movements.
  Arms: Core stability and cognitive training; core stability
Other: Cognitive training — Balance training is combined with a cognitive task involving a backward digit span test, where participants must recall and repeat sequences of numbers in reverse order, testing working memory. This test includes three difficulty levels (3-, 4-, and 5-digit sequences) performed over 35 seconds. Participants will either recall digits while maintaining static stability or after squatting upon hearing a number, with a focus on accuracy within 5 seconds. Performance is measured by the percentage of correctly recalled digits, and error scoring will be documented via video recording for each posture task.
  Arms: Core stability and cognitive training; cognitive training

SUMMARY:
The purpose of the study is to investigate dynamic core stability training versus cognitive training on balance, functional performance, postural control, ankle instability scores, ankle dorsiflexion range of motion, and mental workload in chronic ankle instability

DETAILED DESCRIPTION:
Lateral ankle sprains (LAS) are prevalent in sports, with 40% leading to chronic ankle instability (CAI), impacting muscle coordination and balance, primarily controlled by the central nervous system (CNS). Core muscles play a vital role in stabilization and postural control, particularly for individuals with chronic ankle instability, because they significantly contribute to the risk of injury. Even with intact strength and balance, individuals with chronic ankle instability may re-injure when attention shifts, highlighting the need for dual-task training to improve postural control. Core stability training, which includes cognitive elements, has been shown to enhance muscle function and reduce instability. Training programs incorporating dual-task exercises have proven superior for improving joint position sense and postural control while addressing associated mental health issues in chronic ankle instability patients. Therefore, this study aims to analyze the effects of combining dynamic core stability exercises with cognitive training on dual-task conditions, marking a novel approach in chronic ankle instability rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria will be based on the standard criteria outlined by the International Ankle Consortium

1. History of chronic lateral ankle sprain and/or recurrent sprain and/or "feelings of instability or giving way" for 6 months or more before the study, with at least 2 episodes.
2. Patients are between 18 and 30 years old. 3- Body mass index less than 30

4. The patient has a history of at least one significant ankle sprain with associated inflammatory symptoms and at least one day of interrupted physical activity.

5. Patients who have unilateral chronic ankle instability. 6. Self-reported ankle instability should be confirmed using a validated ankle instability questionnaire (greater than 24).

Exclusion Criteria:

Those with a history of spine, pelvis, and lower extremity injury, fracture, or surgery 2- Those with low back pain that require medical or surgical intervention. 3- Having a history of an acute lower extremity injury or lower extremity surgery or fracture in the 3 months before the Study 4. Participation in formal ankle rehabilitation in the 3 months before the study.

5. Being diagnosed with neurologic dysfunction, such as multiple sclerosis, Parkinson's disease, or head injury

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
assessment of change of pain | at baseline and after 2 months
  Ankle pain will be evaluated using the Arabic version of the Cumberland Ankle Instability Tool, which consists of questions that the patient must answer to reflect their condition. The scoring ranges from 0 to 30, with 0 indicating severe instability and 30 indicating normal stability. A score below 24 suggests Chronic Ankle Instability as defined by the International Ankle Consortium
assessment of ankle instability | at baseline and after 2 months
  Ankle instability will be evaluated using the Arabic version of the Cumberland Ankle Instability Tool, which consists of questions that the patient must answer to reflect their condition. The scoring ranges from 0 to 30, with 0 indicating severe instability and 30 indicating normal stability. A score below 24 suggests Chronic Ankle Instability as defined by the International Ankle Consortium

SECONDARY OUTCOMES:
assessment of foot function | at baseline and after 2 months
  Participants will complete a 29-item questionnaire consisting of the Foot and Ankle Ability Measure, which includes a 21-item Activities of Daily Living (ADL) Subscale and an 8-item Sports Subscale. Each item is rated on a 5-point Likert scale from 0 (unable to perform) to 4 (no difficulty), yielding a potential score of 0 to 84 for the ADL subscale and 0 to 32 for the Sports subscale. The total score is calculated by subtracting the raw score from the maximum possible score, dividing by the maximum score, and multiplying by 100 to determine the percentage of maximum ability achieved.
assessment of functional performance | at baseline and after 2 months
  The side-hop test involves participants hopping laterally on one limb over a distance of 30 cm for 10 repetitions, with a stopwatch recording the fastest time. Trials are invalidated if the contralateral foot touches the ground. After 1-3 practice trials, 3 test trials are conducted, and the average time is used for analysis (Kamonseki et al., 2018). Additionally, the figure of the hop test requires participants to hop twice around a 5-m cone-marked course as fast as possible, with penalties for footfall or course deviations, and timing recorded to the nearest 0.01 seconds.
assessment of postural control | at baseline and after 2 months
  The modified star test grid features three lines emanating from a center point, oriented as anterior, posteromedial, and posterolateral. Participants stand at the center with feet together and perform single-limb squats, reaching towards maximum points along each direction line with the swinging limb. The participant must lightly touch the line with the distal part of the reaching foot without shifting their weight to it or resting on it. They must then return the limb to the center while maintaining balance on the stance limb. Any heavy contact, resting, or shifting during the trial invalidates it. Maximum reach distances are measured with a tape measure.
assessment of balance | at baseline and after 2 months
  The "Self-check" mode provides two measurement options for Static Balance Testing and alternative assessments using an Electronic Balance Board. Participants stand with feet shoulder-width apart (~30 cm) and are monitored via a computer screen displaying a target zone of five concentric circles. The test includes a 15-second adaptation phase followed by a 20-second measurement period, during which stability is assessed based on how long a tracking ball remains within the inner circle. Scores range from 1 (Excellent Stability) to 5 (Bad Stability), with lower scores indicating better performance. Additionally, dynamic tasks require participants to track a target point on-screen, measuring time in the target for scoring. After the tests, scores for each foot and the overall percentage difference are displayed, with values below 10% indicating good body balance.
assessment of Dorsiflexion range of motion | at baseline and after 2 months
  The inclinometer will be fixed to the lateral side of the distal leg just above the ankle joint using a strap. It should be oriented laterally, and its zero point should be parallel to the floor. Participant will make dorsiflexion from weightbearing position by proximal segment, the degree of changed range from zero will be appeared on inclinometer
assessment of mental workload | at baseline and after 2 months
  using the National Aeronautics and Space Administration-Task Load Index questionnaire. Participants assess the workload of a comprehension task after reading selected texts by answering 10 questions. A rater evaluates and assigns weights to six scales based on 15 pair-wise comparisons. Each scale is represented by a line divided into intervals, with descriptors ranging from 'low' to 'high', except for 'performance', which goes from 'good' to 'poor' and is reverse scored. The overall workload score is computed by multiplying raw ratings by participant weights, summing these, and dividing by 15, resulting in a score from 0 to 100.

CONTACTS AND LOCATIONS:
Locations (1):
- out-patient clinic, faculty of physical therapy, Cairo university, Cairo, Egypt